CLINICAL TRIAL: NCT06665893
Title: Evaluating the Efficacy of the Evira Treatment Tool for Childhood Obesity Treatment - a 26- Week Single Arm Interventional Study in Abu Dhabi, United Arab Emirates
Brief Title: Local Proof of Concept of Evira in Abu Dhabi Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Shakhbout Medical City (Other)
Collaborators: Karolinska Institutet (Other); Evira AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EviraUAE
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Childhood Obesity; Adolescent Obesity; Treatment Adherence
Keywords: Digital health; Home-weighing; Obesity treatment; Treatment outcome
MeSH Terms: conditions — Pediatric Obesity; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Children aged 6-15.9 years of age will be asked for participation. Participants included in the study will perform daily weighings at home and parents will be able to follow treatment closely in an application on their phone. Through a communication function in the application, families will be able to communicate in a fast and easy way with healthcare professionals at the clinic. The study duration is 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digi-physical treatment in Abu Dhabi (Experimental): The participants will receive digi-physical treatment using the Evira treatment tool. During the first 2 weeks, participants will receive information about the system and how to utilize the daily weighings and communication system. The families will be informed to perform lifestyle changes that they consider feasible in their specific living situations. The families will get one or two scales, depending on the family situation, and the phone applications installed in the parent's smart phones and, depending on the age of the child, in the child's phone as well. Clinical investigations will be completed and includes physical and abdominal examinations, weight, height, blood pressure and blood sampling. All participants will also be asked to answer questionnaires including quality of life, eating disorders, and treatment satisfaction.
  Interventions: Device: Digi-physical treatment tool

INTERVENTIONS:
Device: Digi-physical treatment tool — A support tool named Evira will be used to provide behavioral treatment. Through daily weightings at home using a special designed scale, which sends data directly to an application on the parents phone and to a clinic homepage, the child's weight development can be easily monitored.

SUMMARY:
Evira is a digital treatment tool developed for treatment of childhood obesity. Through daily weighings at home using a special scale together with a message function in the Evira application, parents and the clinicians can easily follow the child's weight development. The primary aim of this study is to evaluate its efficacy for childhood obesity treatment in Abu Dhabi, with a secondary objective to establish non-inferiority compared to outcomes in a cohort in Stockholm, Sweden.

DETAILED DESCRIPTION:
Obesity remains a critical global health concern. Traditional treatment often yields limited results, necessitating innovative solutions.

In this study, participants aged 6-15.9 years with obesity at the Sheikh Shakabout Medical City in Abu Dhabi, will be asked for participation. If agreed to participate, they will use a digital treatment tool as a complement to behavioral treatment.The treatment is based on outcome goals set by the treatment staff together with the family. Briefly, the families follow the child's weight outcome via daily weight measurements and the outcome is shown graphically in the mobile application as BMI SDS with the BMI SDS weight goals as background. The staff will provide support to the families via the app. The staff is encouraged to react and contact the families if the weight goals are not reached or if they fail to perform the daily weighings. Regular physical visits at baseline, 3 months, and 6 months, alongside questionnaire assessments, will facilitate data collection via electronic case report forms.

The purpose of this study is to evaluate the treatment tools efficacy for childhood obesity treatment in Abu Dhabi. Furthermore, the study aims to establish non-inferiority compared to outcomes in Stockholm, Sweden (referred to as the "Stockholm cohort"), on 107 children and adolescents who were treated with the same treatment method between October 2018 and August 2019 (Clinicaltrials.gov ID: NCT04323215).

ELIGIBILITY:
Inclusion Criteria:

* Age >6.0 and <16.0 years of age at inclusion
* Obesity according to International Obesity Task Force (IOTF)
* Willingness to participate in an obesity treatment proof of concept trial
* Family ability to communicate e.g. write and read messages in the mobile application
* Parents having a smart phone and an email address

Exclusion Criteria:

* Morbid obesity defined as iso-BMI>40 kg/m2 independently of age
* Endocrine disorders other than well controlled hypothyroidism
* Metabolic disorders of importance for weight control
* Treatment for depression and other psychiatric disorders during the last 6 months before inclusion
* Pharmacological treatment of importance for weight control
* Hypothalamic or monogenic obesity, e.g. syndromes and Mb Down
* Severe neuropsychiatric disorders that could affect study compliance
* Eating disorders requiring therapy during the last six months before inclusion or observed at the inclusion screening.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in degree of obesity | From start of treatment to six months follow-up
  Measured by BMI standard deviation score.

SECONDARY OUTCOMES:
Proportion of individuals reaching a clinically significant change in relative weight | From start of treatment to six months follow-up
  Proportion of individuals reaching a clinically significant change in relative weight defined as a decrease of -0.20 BMI SDS units. Abu Dhabi cohort vs. Stockholm cohort
Proportion of individuals in obesity remission | From start of treatment to six months follow-up
  Obesity remission defined as no longer having obesity class 1. Abu Dhabi cohort vs. Stockholm cohort
The use of the support tool - weighings | From start of treatment to six months follow-up
  Number of weighings/week. Abu Dhabi cohort vs. Stockholm cohort
The use of the support tool - text messages | From start of treatment to six months follow-up
  Number of weighings/week. Abu Dhabi cohort vs. Stockholm cohort
Number of physical visits | From start of treatment to six months follow-up
  Visits to the clinic. Abu Dhabi cohort vs. Stockholm cohort
Number of cancelation of physical visits | From start of treatment to six months follow-up
  Visits to the clinic. Abu Dhabi cohort vs. Stockholm cohort
Number of patients not showing up to physical visits | From start of treatment to six months follow-up
  Visits to the clinic. Abu Dhabi cohort vs. Stockholm cohort
Psycho-social health measures | From start of treatment to six months follow-up
  Psycho-social health assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire. The PROMIS questionnaire is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The output from a PROMIS score is represented as a T score. Higher scores indicate more of the domain being measured (e.g., more fatigue, more pain).
Drop-out rate | From start of treatment to six months follow-up
  Number of drop-outs. Abu Dhabi cohort vs. Stockholm cohort
Change in degree of obesity. Abu Dhabi cohort vs. Stockholm cohort | From start of treatment to six months follow-up
  Measured by BMI standard deviation score

CONTACTS AND LOCATIONS:
Overall Officials: Asma Deeb, Dr., Principal Investigator — Sheikh Shakhbout Medical City Abu Dhabi
Locations (1):
- Sheikh Shakhbout Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for the main outcome will be available upon date of scientific publications. To preserve individual case and anonymity, more detailed data and additional variables will be available upon request.